CLINICAL TRIAL: NCT00763230
Title: A Sham-controlled Study of Transcranial Direct Current Stimulation (tDCS) as a Treatment for Depression
Brief Title: A Study of Transcranial Direct Current Stimulation (tDCS) to Treat Depression
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of New South Wales (Other)
Responsible Party: Associate Professor Colleen Loo, University of New South Wales
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07305; NHMRC (Australia)
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2011-03

CONDITIONS: Depressive Disorder, Major; Bipolar Disorder
Keywords: Depression; Treatment; Transcranial direct current stimulation
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Depression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- active (Experimental): Full active tDCS treatment
  Interventions: Device: Transcranial direct current stimulation
- sham (Sham Comparator): Placebo tDCS will be give
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — tDCS will be given every weekday. For each session, tDCS will be given continuously for 20 minutes at 2 mA. Conductive rubber electrodes (7 x 5 cm, 35 cm2) covered by sponges soaked in saline will be used, held in place by a head band. The current will be gradually increased to the level of 2 mA over 30 seconds (to avoid the sensation of a flash as described in the safety section above). For sham stimulation, the current will be left on for another 30s, then gradually reduced to zero over another 30 seconds, so that the initial tingling sensation experienced by subjects will be identical for the two groups. The stimulator will be placed behind the subject's head so any adjustments to the current by the operator are not evident. This sham procedure resulted in successful blinding in our pilot study.
  Other Names: Eldith DC-Stimulator (CE certified)

SUMMARY:
Depression is a common illness with an approximate lifetime prevalence of 17 %, conferring a large burden of disease in the community, often due to inadequate treatment. Thus there is interest in the therapeutic potential of non invasive, novel forms of brain stimulation, such as transcranial direct current stimulation (tDCS). Two small studies have been published in the last two years indicating that 20 minutes of either 1 or 2mA tDCS over 5 or 10 sessions is safe, painless and well tolerated. The investigators' own pilot data (N=30) also suggests the technique has antidepressant effects and is safe (5-10 sessions of tDCS at 1 mA).

This study will extend previous findings, testing a more definitive tDCS approach (also left prefrontal anodal stimulation) with a longer treatment course (15 sessions), at 2 mA (which has been found to be safe and more effective than 1 mA in cognitive studies), and in a larger sample (N=68), using a placebo-controlled design.

It is hypothesised that active tDCS (15 sessions) will have greater efficacy than sham treatment (15 sessions) in reducing the severity of depressive symptoms in patients in an episode of major depression. A second hypothesis is that 15 sessions of tDCS will not cause any significant adverse effects or cause decline in neuropsychological functioning in comparison to a sham control.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for DSM-IV Major Depressive Episode

Exclusion Criteria:

* Diagnosis (as defined by DSM-IV) of: any psychotic disorder except bipolar disorder(lifetime); eating disorder (current or within the past year); obsessive compulsive disorder (lifetime); post-traumatic stress disorder (current or within the past year); mental retardation.
* History of drug or alcohol abuse or dependence (as per DSM-IV criteria) within the last 3 months (except nicotine and caffeine).
* Inadequate response to ECT in the current episode of depression.
* Subject is on regular benzodiazepine medication which it is not clinically appropriate to discontinue.
* Subject requires a rapid clinical response due to inanition, psychosis or high suicide risk.
* Neurological disorder or insult, eg recent stroke (CVA), which places subject at risk of seizure or neuronal damage with tDCS.
* Subject has metal in the cranium, skull defects, or skin lesions on scalp (cuts, abrasions, rash) at proposed electrode sites.
* Female subject who is pregnant, or of child-bearing age, sexually active and not using reliable contraception

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2008-04; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale for Depression (MADRS) | 6 months
  Baseline (pre-treatment), post 8, 15, 23 and 30 tDCS sessions, and follow-up 1 week, 1 month, 3 months and 6 months post treatment

SECONDARY OUTCOMES:
Inventory of Depressive Symptomatology (IDS-C) | 6 months
  Baseline (pre-treatment), post 8, 15, 23 and 30 tDCS sessions, and follow-up 1 week, 1 month, 3 months and 6 months post treatment
Quick Inventory of Depressive Symptomatology - Self rated (QIDS-SR) | Baseline (pre-treatment), post 8, 15, 23 and 30 tDCS sessions, and follow-up 1 week, 1 month, 3 months and 6 months post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Loo, Principal Investigator — University of New South Wales
Locations (1):
- Black Dog Institute, University of New South Wales, Randwick, New South Wales, Australia

REFERENCES:
- [Derived] Loo CK, Alonzo A, Martin D, Mitchell PB, Galvez V, Sachdev P. Transcranial direct current stimulation for depression: 3-week, randomised, sham-controlled trial. Br J Psychiatry. 2012 Jan;200(1):52-9. doi: 10.1192/bjp.bp.111.097634. PMID 22215866
- See also: Black Dog Institute website — http://www.blackdoginstitute.org.au